CLINICAL TRIAL: NCT07291167
Title: Study on the Correlation Between Metabolomics and Anxiety and Depression in Bronchiectasis
Status: Not yet recruiting | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Wang xiaorong, Internal medicine physician, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: 2025XHHX001
Record Dates: First submitted 2025-09-25; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Bronchiectasis
Keywords: Bronchiectasis; Depression; Anxiety
MeSH Terms: conditions — Bronchiectasis; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, sputum, stool would be collected and stored at - 80℃
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: inapplicable — This study is observational in nature and did not involve any intervention measures.

SUMMARY:
Bronchiectasis is a common lung disease. Approximately 20-40% of patients with bronchiectasis experience comorbid anxiety and depression. Multiple studies have now demonstrated that anxiety and depression are associated with an increased risk of disease exacerbation in these individuals.

Therefore, this study aims to collect data on anxiety and depression status, disease exacerbation frequency, hospitalisation rates, and mortality among participants diagnosed with bronchiectasis. Concurrently, biological samples including blood, sputum, and stool will be obtained. Through metabolomics analysis, we will investigate the expression of anxiety and depression-related metabolic pathways and identify corresponding biomarkers to explore their role in the progression of bronchiectasis.

DETAILED DESCRIPTION:
Non-cystic fibrosis bronchiectasis is a common pulmonary disorder. Recurrent acute exacerbations of bronchiectasis can severely impair lung function, accelerate the decline of pulmonary capacity, diminish quality of life and shorten survival duration. While previous studies have identified factors such as deteriorating lung function and Pseudomonas aeruginosa infection as contributing to acute exacerbations, eliminating these factors does not entirely prevent such episodes in patients with bronchiectasis. Current research suggests that 20-40% of patients with bronchiectasis experience anxiety and/or depression. These conditions are associated with an increased risk of disease exacerbation, with depression specifically linked to a shorter time to first exacerbation. Therefore, investigating the intrinsic role of anxiety and depression in disease progression is crucial.

According to the inclusion and exclusion criteria, this study will enroll participants diagnosed with bronchiectasis at Union Hospital, Tongji Medical College of Huazhong University of Science and Technology, Guizhou Provincial People's Hospital, and Yichang Central Hospital between December 20, 2025, and December 31, 2030. The study protocol was approved by the research ethics boards at each hospital. At enrolment, the following demographic information will be collected: gender, age, height (in metres) and weight (in kilograms). Medical history, previous exacerbations and blood test results (including complete blood count and biochemical parameters) will also be obtained during the initial consultation. Pathogenic examination results will also be recorded. Additionally, pulmonary function tests (e.g. FEV1% predicted) and high-resolution computed tomography (HRCT) scans of the lungs will be performed. Patients' breathlessness will be assessed using the modified Medical Research Council (mMRC) dyspnoea scale, while anxiety and depression status will be evaluated using the Hospital Anxiety and Depression Scale (HADS). With informed consent, biological samples, including blood, sputum and stool, were collected. Participants underwent follow-up every three months post-enrolment, with records maintained of exacerbation frequency, hospitalisation episodes and survival status. Upon completion of data collection, metabolomic analysis will be performed on samples including blood, sputum, and stool to investigate whether patients' anxiety and depression states are associated with the aforementioned metabolomic findings, identify corresponding biomarkers, and analyze the role of anxiety and depression in the progression of bronchiectasis.

Materials and Methods

1. Data Collection Inclusion and exclusion criteria

   Inclusion Criteria:
   * Age ≥18 years
   * Participants' pulmonary imaging findings and clinical presentation met the diagnostic criteria for bronchiectasis
   * Clinically stable (no antibiotics or oral corticosteroids within 4 weeks prior to enrolment);
   * Patients who are willing to sign the consent form and participate in the study.

   Exclusion Criteria:
   * Age <18 years
   * Does not meet the diagnostic criteria for bronchiectasis
   * Participants with cystic fibrosis or previous lung transplantation
   * Participants who are unable to cooperate with the study due to dysfunction of vital systems such as heart, brain, liver, and kidneys, or who are unable to participate in the study due to comorbid serious diseases
   * Participants with active disorders, including active tuberculosis, active allergic bronchopulmonary aspergillosis, active nontuberculous mycobacterial infection and malignancy or secondary traction bronchiectasis associated with pulmonary fibrosis
   * Pregnant or lactating females
   * Who are not able to provide informed consent or who refuse to participate in the clinical study

   Collection of patient demographic indicators and laboratory test results. Demographic indicators (age, height, weight), mMRC score, laboratory test results, pulmonary function (FEV1% predicted), radiological scores (modified Reiff, Bhalla score) were collected upon participant enrolment.

   Assessment of Anxiety and Depression Status：All patients were requested to complete the Hospital Anxiety and Depression Scale (HADS) at baseline. The score for each subscale (HADS depression and anxiety) ranges from 0 to 21 points, with a score ⩾8 indicating probable depression or anxiety .

   Assessment of Disease Severity：Disease severity was evaluated using the Bronchiectasis Severity Index (BSI).
2. Metabolomics Experimental MethodsMetabolomics Experimental Methods 2.1 Sample Preparation 50 μL of collected sample was thawed on ice and mixed with 200 μL of cold methanol:acetonitrile (1:1, v/v) containing the IS (1 μg/mL). The mixture was vortexed vigorously, incubated at -20°C for 2 h, and then centrifuged at 14,000 g for 15 min at 4°C. The supernatant was transferred to a new vial for LC-MS analysis. A pooled quality control (QC) sample was prepared by combining equal aliquots from all individual samples.

   2.2 LC-MS Analysis Chromatographic separation was performed on a Waters ACQUITY UPLC system using a HSS T3 column (2.1 × 100 mm, 1.8 μm) maintained at 40°C. The mobile phase consisted of (A) water with 0.1% formic acid and (B) acetonitrile with 0.1% formic acid. A linear gradient was applied as follows: 0-2 min, 2% B; 2-10 min, 2% to 98% B; 10-12 min, 98% B; 12-12.1 min, 98% to 2% B; 12.1-15 min, 2% B. The flow rate was 0.4 mL/min and the injection volume was 2 μL.

   > Mass spectrometry was conducted on a SCIEX TripleTOF 6600+ system operated in both positive and negative ESI modes. The parameters were set as follows: Ion Source Gas 1: 60 psi, Ion Source Gas 2: 60 psi, Curtain Gas: 35 psi, Source Temperature: 550°C, Ion Spray Voltage: ±5500 V. Data were acquired in information-dependent acquisition (IDA) mode.

   2.3 Data Processing and Multivariate Statistical Analysis Raw data files were processed using MS-DIAL software for peak picking, alignment, and normalization against the IS. The resulting data matrix was imported into SIMCA-P software (v16.0, Umetrics, Sweden) for multivariate analysis. Unit variance scaling and mean centering were applied prior to PCA and OPLS-DA. The OPLS-DA model was validated by a 200-time permutation test.

   Metabolites with Variable Importance in Projection (VIP) > 1.0 from the OPLS-DA model and p-value < 0.05 from univariate Student's t-test were considered statistically significant.

   2.4 Metabolite Identification Significant metabolites were identified by comparing their accurate mass (mass error < 10 ppm) and MS/MS spectra with entries in the HMDB database. Where possible, identification was confirmed by comparison with authentic standards (Level 1 confidence).
3. Clinical Data Statistical Analysis and Methods:

The data obtained during the study were pre-collated. For continuous data, normality tests were first performed. If all groups met normality, the Student's t-test was used for comparison between groups. Otherwise, the non-parametric Wilcoxon rank sum test was considered. For categorical variables, the χ2 test was used. Statistically significant data were subjected to multivariate logistic regression analysis. P < 0.05 was deemed statistically significant.

Statistical analysis of all data was performed through SPSS (IBM SPSS Statistics 26.0, SPSS Inc., Chicago, IL) and R language (version 4.1.3, www.R-project.org/). All statistical tests were two-sided, and statistical significance was set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Participants' pulmonary imaging findings and clinical presentation met the diagnostic criteria for bronchiectasis
* Clinically stable (no antibiotics or oral corticosteroids within 4 weeks prior to enrolment);
* Patients who are willing to sign the consent form and participate in the study.

Exclusion Criteria:

* Age <18 years
* Does not meet the diagnostic criteria for bronchiectasis
* Participants with cystic fibrosis or previous lung transplantation
* Participants who are unable to cooperate with the study due to dysfunction of vital systems such as heart, brain, liver, and kidneys, or who are unable to participate in the study due to comorbid serious diseases
* Participants with active disorders, including active tuberculosis, active allergic bronchopulmonary aspergillosis, active nontuberculous mycobacterial infection and malignancy or secondary traction bronchiectasis associated with pulmonary fibrosis
* Pregnant or lactating females
* Who are not able to provide informed consent or who refuse to participate in the clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with all-cause bronchiectasis would be included, such as those with tuberculosis history and genetic disorders.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of acute exacerbations of bronchiectasis | up to 5 years
  Acute exacerbations of bronchiectasis were defined according to the consensus published in the European Journal of Respiratory Sciences in 2017, and the frequency of acute exacerbations per year was obtained from participants through follow-up visits

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | Lasts for 5 years
  Assess the patient using the Hospital Anxiety and Depression Scale (HADS), and record the information at least once a year for a duration of 5 years.
Lung Function FVC measured in liters (L) | recorded at baseline and re-tested every year, up to 5 years.
Lung Function FEV1% | recorded at baseline and re-tested every year, up to 5 years.
Lung Function - The FEV1/FVC ratio | recorded at baseline and re-tested every year, up to 5 years.
modified Medical Research Council (mMRC) dyspnea score | At baseline and updated once a year for 5 years
  The mMRC score primarily assesses the degree of a patient's chest tightness, shortness of breath, and difficulty breathing during various levels of physical activity.
Bhalla scores on CT of participants' lungs | Assess once a year from the start of enrollment, for a total duration of five years.
  A Bhalla severity score was performed and recorded on lung CT at enrolment and during annual follow-up. The Bhalla score is 0-25, with higher scores indicating greater severity.
Frequency of hospitalisation | Starting from inclusion in the study, data will be summarized once per year for a total duration of five years.
  Frequency of hospitalisation for bronchiectasis among participants in a year
Mortality rate | Five-year mortality rate
  Participants died during follow-up because of bronchiectasis as the main cause of death.
Bronchiectasis severity Score (BSI) | At baseline and updated once a year for 5 years
  The scale is presented online. It consists of 9 items including Age, BMI(Body Mass Index), % FEV1 Predicted, Previous Hospital Admission in the past 2 years, number of exacerbations in previous year, MRC Breathlessness Score, Pseudomonas Colonisation, Colonisation with other organisms,affected lobes.
  0-4 Mild Bronchiectasis. 5 - 8 Moderate Bronchiectasis. 9 + Severe Bronchiectasis.
E-FACED score | At baseline and updated once a year for 5 years
  It consists of 6 items including exacerbation history in the past year, % FEV1 predicted, Age, Chronic colonization by Pseudomonas aeruginosa, n° of pulmonary lobes affected,and Dyspnea (measured by mMRC score) mild: 0-3 points, moderate: 4-6 points; and severe: 7-9 points
Quality of Life Questionnaire-Bronchiectasis | At baseline and updated once a year for 5 years
  The questionnaire asks patients questions about their current state of health. It could be downloaded from the website online.
Microbiology checklist | At least 1 year before enrollment and 5 years during the follow-up
  Microorganisms cultured from sputum or bronchoalveolar lavage fluid

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Union Hospital,China, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
In this study, we will share parts of the study design such as Study Protocol, Statistical Analysis Plan (SAP) and Informed Consent Form (ICF).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: We will share the data 6 months after the end of the study, which lasts for 3 years
Access Criteria: Data were obtained through the Principal Investigator of this study upon reasonable request.

REFERENCES:
- [Result] Polverino E, Goeminne PC, McDonnell MJ, Aliberti S, Marshall SE, Loebinger MR, Murris M, Canton R, Torres A, Dimakou K, De Soyza A, Hill AT, Haworth CS, Vendrell M, Ringshausen FC, Subotic D, Wilson R, Vilaro J, Stallberg B, Welte T, Rohde G, Blasi F, Elborn S, Almagro M, Timothy A, Ruddy T, Tonia T, Rigau D, Chalmers JD. European Respiratory Society guidelines for the management of adult bronchiectasis. Eur Respir J. 2017 Sep 9;50(3):1700629. doi: 10.1183/13993003.00629-2017. Print 2017 Sep. PMID 28889110
- [Result] Hill AT, Sullivan AL, Chalmers JD, De Soyza A, Elborn SJ, Floto AR, Grillo L, Gruffydd-Jones K, Harvey A, Haworth CS, Hiscocks E, Hurst JR, Johnson C, Kelleher PW, Bedi P, Payne K, Saleh H, Screaton NJ, Smith M, Tunney M, Whitters D, Wilson R, Loebinger MR. British Thoracic Society Guideline for bronchiectasis in adults. Thorax. 2019 Jan;74(Suppl 1):1-69. doi: 10.1136/thoraxjnl-2018-212463. No abstract available. PMID 30545985
- [Result] Lee JH, Lee WY, Yong SJ, Kim WJ, Sin S, Lee CY, Kim Y, Jung JY, Kim SH; KMBARC. Prevalence of depression and its associated factors in bronchiectasis: findings from KMBARC registry. BMC Pulm Med. 2021 Sep 27;21(1):306. doi: 10.1186/s12890-021-01675-4. PMID 34579692
- [Result] Gao YH, Guan WJ, Zhu YN, Chen RC, Zhang GJ. Anxiety and depression in adult outpatients with bronchiectasis: Associations with disease severity and health-related quality of life. Clin Respir J. 2018 Apr;12(4):1485-1494. doi: 10.1111/crj.12695. Epub 2017 Sep 19. PMID 28842946
- [Result] Gao YH, Zheng HZ, Lu HW, Li YY, Feng Y, Mao B, Bai JW, Liang S, Cheng KB, Gu SY, Sun XL, Li JX, Ge A, Li MH, Yang JW, Bai L, Yu HY, Qu JM, Xu JF. The impact of depression and anxiety on the risk of exacerbation in adults with bronchiectasis: a prospective cohort study. Eur Respir J. 2023 Feb 2;61(2):2201695. doi: 10.1183/13993003.01695-2022. Print 2023 Feb. No abstract available. PMID 36669778